CLINICAL TRIAL: NCT00013923
Title: A Nutritional Brain Metabolic Enhancer for Alzheimer Disease
Brief Title: Effectiveness of A Nutritional Brain Metabolic Enhancer for Alzheimer Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Burke Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA0027
Record Dates: First submitted 2001-04-02; First posted 2001-04-03 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2003-08

CONDITIONS: Alzheimer Disease
Keywords: Nutritional Supplement
MeSH Terms: conditions — Alzheimer Disease | interventions — Dietary Supplements

INTERVENTIONS:
Drug: Nutritional Supplement

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a nutritional supplement that has been developed to improve the brain function of a patient with Alzheimer's disease.

DETAILED DESCRIPTION:
The ability of the brain to use its major fuel, the sugar glucose, is reduced in Alzheimer's disease. A nutritional supplement has been developed to improve the function of the Alzheimer brain by increasing its ability to use sugar effectively. The ingredients of the supplement are natural products, and are found in the normal American diet. Results have been encouraging in open trials where the patients knew they were taking the active medicine. Patients are now being invited to participate in a placebo-controlled trial lasting 3 months, followed by a 3-month open label trial where all patients will receive the active preparation.

This is a double-blind, placebo-controlled, parallel-group, 3 month trial followed by a 3-month open-label period, of a nutritional supplement designed to improve brain metabolism and function in patients with Alzheimer's disease (AD). The design of the nutritional supplement is based on replicated observations of abnormalities in mitochondria in AD. The constituents of the nutritional supplement are components of the normal American diet, and are classified by the FDA as GRAS (Generally Regarded As Safe). Results with the supplement have been favorable in preliminary, open trials (eg mean improvement in MMSE score of +4.9, range +3 to +8, n = 7, P <0.0004).

During the placebo-controlled portion of the trial, half of the participants will receive the active preparation and half a sugar pill. During this first phase, neither the patients nor those testing them will know who is taking active medicine and who is taking placebo. The active supplement or placebo are taken as 1 tablespoon twice a day, between meals. If desired, the supplement or placebo can be stirred into, or washed down with, water, coffee or tea without milk or sugar, or the soft drink TAB. Patient visits to the Burke Medical Research Institute will be once a month, after the screening and baseline visits.

The supplement is taken as one tablespoon of a fluid, between meals. Since other sugars or citrate can be expected to interfere with the actions of the supplements, food or drinks containing sugar or citrate and diet drinks containing citrate are to be avoided for 1 1/2 hour before and 1 1/2 hour after taking the supplement. No significant adverse events have been associated with this supplement. However, standard precautions for patient safety are being taken, including medical examination and clinical laboratory tests at screening and at the completion of the double-blind and open-label phases.

ELIGIBILITY:
Inclusion criteria include:

* A documented diagnosis of Alzheimer's disease;
* MMSE score between 10 and 26 inclusive;
* A reliable caregiver to ensure compliance.

Exclusion criteria include:

* diabetes, unstable medical illness, myocardial infarction or cancer diagnosed within the previous 12 months, or treatment with systemic steroids.
* Patients being treated for depression or other psychiatric symptomatology are eligible, if their symptoms are under control on a stable dose of medication

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Blass, MD, PhD, Principal Investigator — Burke Medical Research Institute
Locations (1):
- Burke Medical Research Institute, White Plains, New York, United States

REFERENCES:
- [Background] Blass JP. The mitochondrial spiral. An adequate cause of dementia in the Alzheimer's syndrome. Ann N Y Acad Sci. 2000;924:170-83. doi: 10.1111/j.1749-6632.2000.tb05576.x. PMID 11193795
- [Background] Blass JP, Sheu RK, Gibson GE. Inherent abnormalities in energy metabolism in Alzheimer disease. Interaction with cerebrovascular compromise. Ann N Y Acad Sci. 2000 Apr;903:204-21. doi: 10.1111/j.1749-6632.2000.tb06370.x. PMID 10818509
- [Background] Manning CA, Ragozzino ME, Gold PE. Glucose enhancement of memory in patients with probable senile dementia of the Alzheimer's type. Neurobiol Aging. 1993 Nov-Dec;14(6):523-8. doi: 10.1016/0197-4580(93)90034-9. PMID 8295654